CLINICAL TRIAL: NCT00836394
Title: The Effect of Whole Body Vibration Therapy on Muscle Function and Joint Loading in Children With Juvenile Idiopathic Arthritis
Brief Title: Effect of Whole Body Vibration Therapy in Children With Juvenile Idiopathic Arthritis
Acronym: WBV-JIA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No potential participants met entry criteria
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Canadian Arthritis Network (Network); University of Ottawa (Other)
Responsible Party: Principal Investigator, Johannes Roth, MD, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBV-JIA
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: arthritis; juvenile idiopathic arthritis; pediatric; intervention; vibration therapy; JIA
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Will undergo whole body vibration (WBV) therapy (6 minutes of training on 5 days a week for 3 months)
  Interventions: Device: Galileo (whole body vibration (WBV) therapy)
- Control (No Intervention): Will follow daily habitual activities

INTERVENTIONS:
Device: Galileo (whole body vibration (WBV) therapy) — 6 minutes of training on 5 days a week for 3 months
  Other Names: Galileo
  Arms: Intervention Group

SUMMARY:
Juvenile idiopathic arthritis (JIA) is one of the most common chronic illnesses in children, with recent data suggesting that 1 to 4 in 1000 Canadian children and youth cope with the condition. Many JIA children will enter adulthood with permanent joint damage5. In parallel, a significant number are affected by deficits of muscle function. In addition to the impact on physical function, muscles play an important role in maintaining joint health. The overall aim of this proposal is to evaluate a novel therapeutic intervention - whole body vibration (WBV) - for its ability to improve muscle function and the biomechanics of lower extremity joints in JIA in order to prevent joint degeneration.

DETAILED DESCRIPTION:
This project aims to evaluate the effect of a therapy called whole body vibration (WBV) on muscle function and joint biomechanics in children and adolescents suffering from juvenile idiopathic arthritis (JIA).

JIA is the most common chronic form of arthritis in children and affects at least 1 in 1000 Canadian children and youth. Current data suggests that a large number of children suffering from JIA will encounter permanent joint damage, to which direct effects of inflammation are an important contributor. Nevertheless, recent research has also shown that impaired muscle function and a subsequent alteration of joint loading might by itself induce joint damage. Fifty percent of JIA patients have significant impairments of muscle function and this is often present in patients who do not have active arthritis anymore. In addition to optimum medical treatment of the disease, it is therefore important to improve muscle function in order to protect the joints.

WBV therapy might be an interesting technique to achieve this in JIA patients. It is able to improve muscle function very efficiently with relatively short training times and at the same time confers loads to the lower limbs which are only 30% of body weight. The WBV device consists of a plate going up and down along a fulcrum at a high frequency. The patient stands on the WBV device and the vibration will induce muscle stretch reflexes producing muscle contractions. These muscle contractions are similar to muscle activity during exercise and are not perceived as painful or unpleasant. The technique has been used in children with several conditions impairing muscle function.

The primary question to be investigated in the proposed study is whether WBV therapy will significantly improve muscle function in JIA patients. In addition, the effect of an improvement in muscle function on gait and the loading of individual joints at the lower extremity will be examined. Finally the effect of WBV therapy on quality of life will be assessed.

We propose conducting a controlled trial investigation. This implies, that one group of study participants, called the intervention group, will do the WBV therapy, whereas a second group, called the control group, will just follow their daily habitual activities. All participants will have an initial assessment of muscle function, electrical muscle activity and joint biomechanics by completely painless measurement techniques at the Children's Hospital of Eastern Ontario (CHEO) and a nearby Human Motion Biomechanics lab at the University of Ottawa. In addition, an MRI of the lower legs without contrast media will be done to confirm the absence of joint effusions as well as bone or muscle edema. Quality of life will be assessed by a standard questionnaire that has been validated in JIA. Subsequently, study participants in the intervention group as well as their parents will be introduced to the therapy during two separate sessions at the CHEO. They will then take a WBV device home and perform 6 minutes of training on 5 days a week for 3 months. Each month, they will return to CHEO for assessment of muscle function and demonstration of training technique. At the end of the 3 month period, both intervention and control group patients will repeat the initial set of assessments including MRI. After another 3 month period, all participants will return for a final assessment of muscle function and joint biomechanics but not MRI to document persistence of any change observed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of JIA
* No active lower-limb arthritis at recruitment shown by clinical examination or MRI
* No active arthritis in the 3 months prior to study entry
* Age > 7 years and < 18 years
* Written informed consent from parents and patients over 14 years of age, assent from children 7 to 14 years
* Written commitment by parents to supervise each therapy session
* Z-score power ≤ -1 as determined on the Leonardo force plate

Exclusion Criteria:

* Lower-limb arthritis on clinical examination or MRI
* Acute venous thrombosis
* Acute hernia
* Migraine
* Epilepsy
* Pregnancy
* Participation in another interventional study
* Surgery and/or fracture within previous 3 months
* Joint replacements

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the effect of whole body vibration therapy on muscle function by measuring the increase in z-score muscle power during a two leg jump as determined by jumping mechanography after 12 weeks compared to baseline. | 12 weeks

SECONDARY OUTCOMES:
The increase in muscle force measured during a one leg jump as determined by jumping mechanography | 12 weeks
The increase in joint moment and power of the lower-limb measured in a gait lab using motion analysis | 12 weeks
The change in range of motion, velocity and step distance during walking measured by motion analysis and on the Leonardo gangway | 12 weeks
Muscle activation changes in amplitude and frequency content measured by surface EMG | 12 weeks
The safety of the therapy by documenting any recurrence of joint effusions, bone marrow or muscle edema as determined by MRI imaging of the lower extremity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Roth, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada